CLINICAL TRIAL: NCT06327282
Title: the Effect of Preoperative Pain Education by Anesthesia Nurses on Postoperative Pain Among Adult Patients Undergoing Abdominal Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Hao Li, associate chief physician, Chinese PLA General Hospital
Other Study IDs: ChinaPLAGHPAIN
Record Dates: First submitted 2024-03-17; First posted 2024-03-25 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intervention group: Anesthesia nurses carried out pain-related knowledge education.
  Interventions: Behavioral: education on pain and related knowledge
- Blank group: Patients who did not receive any knowledge education.

INTERVENTIONS:
Behavioral: education on pain and related knowledge — Before surgery, pain related knowledge was educated.
  Other Names: pain-related knowledge education
  Groups: Intervention group

SUMMARY:
To explore the effects of preoperative pain education on postoperative pain among patients undergoing abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

1. voluntary informed consent;
2. age older than 18 years
3. abdominal surgery under elective general anesthesia

Exclusion Criteria:

1. Patients taking long-term analgesics (including opioids, non-steroids, etc.)
2. Patients with preoperative chronic pain
3. Have participated in clinical studies in other projects within 3 months prior to signing the informed consent form
4. subjects not considered by the investigator
5. subjects refused to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing Abdominal Surgery
Sampling Method: Probability Sample
Enrollment: 116 (Estimated)
Dates: Start 2024-06-15 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-04-04 (Estimated)

PRIMARY OUTCOMES:
Occurrence of pain | The first day to the fifth day after surgery.
  The NRS scale was used to evaluate the scores.

SECONDARY OUTCOMES:
Mastery of the use of patient-controlled analgesia pump | Day 2 after surgery
  A series of questions were used to assess patients' mastery of patient-controlled analgesia pump use.

OTHER OUTCOMES:
Patient satisfaction with postoperative analgesia | Day 5 after surgery
  Patient satisfaction with postoperative analgesia
Adverse events of patients using analgesic pump were recorded | The first day to the fifth day after surgery.
  Nausea and vomiting, itching, drowsiness, dizziness
The number of times that the analgesic pump was pressed during each 24h and the amount of analgesic pump remaining at this time were recorded | The first to three days after surgery
  The number of times that the analgesic pump was pressed during each 24h and the amount of analgesic pump remaining at this time were recorded
The use of rescue analgesics after surgery | The first day to the fifth day after surgery.
  Temporary painkillers used in the ward
The postoperative sleep status of patients was evaluated | The first day to the fifth day after surgery.
  The Richards-Campbell Sleep Questionaire Scale was used

IPD SHARING:
Plan to Share IPD: No